CLINICAL TRIAL: NCT04215900
Title: The Impact of High-speed Yoga on Executive Function and Functional Ability in Individuals Diagnosed With Parkinson's Disease.
Brief Title: High-Speed Yoga and Executive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20191202
Record Dates: First submitted 2019-12-10; First posted 2020-01-02 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Executive Dysfunction; Parkinson Disease; Quality of Life
Keywords: Exercise Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Speed Multi-Directional Yoga (Experimental): The duration of the intervention is 18 weeks, with 16 weeks of training.
  Interventions: Behavioral: High-speed yoga multi-directional yoga
- Waitlist control (No Intervention): During the course of the 18 week study this arm will receive no intervention. Participants will be encouraged to maintain their daily schedules.Following the completion of the study the participants will be offered eight yoga sessions over a one month period.

INTERVENTIONS:
Behavioral: High-speed yoga multi-directional yoga — The yoga training will be performed over a 4-month period where classes will be held two times per week. Each session will include a warm-up, speed and balance training section, and cooldown phase. The yoga program will include four separate progressions with the first four weeks serving as a familiarization phase, where the participants will be introduced to the poses and proper technique will be demonstrated. The second four-week phase will emphasize a speed component used to target improvements in aerobic capacity. The same poses previously learned will be used. The final two phases will increase in intensity maintaining the speed element and include skill-based training, where the participants will be asked to complete each pose moving as quickly as possible in response to visual and auditory cues.
  Arms: High-Speed Multi-Directional Yoga

SUMMARY:
The purpose of this research study is to establish if a novel high-speed yoga program which incorporates visual cues can make a positive change in the participant's ability to make decisions and move as measured by several cognitive, balance and functional tests. It has been shown that yoga can improve balance and movement in those diagnosed with Parkinson's disease.

DETAILED DESCRIPTION:
The purpose of this research study is to establish if a novel high-speed yoga program which incorporates visual cues can make a positive change in the participant's ability to make decisions and move as measured by several cognitive, balance and functional tests. It has been shown that yoga can improve balance and movement in those diagnosed with Parkinson's disease. Subjects will be randomly assigned to either the high-speed yoga group or an inactive control group. All subjects will be tested before and after the 16 week training period using tests of balance, cognition and functional movement. The high-speed yoga group will receive yoga sequences lead by a certified yoga instructor during each of the 32 visits to the yoga studio. Each session will last one hour and be conducted two times per week. The program will consist of several different balance poses and movements where participants are encouraged to move quickly. Participants will also be asked to move in different directions based on colored lines placed on the yoga mat. To ensure a safe environment, several assistants will be present to help participants move into each pose. In addition, several assistive devices such as chairs and yoga blocks will be available if participants chose to use them.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 50 and 85 years of age (inclusive);
2. Diagnosis of Parkinson's Disease (Hoehn and Yahr scale I-III);
3. Ability to ambulate with or without an assistive device for at least 50 ft;
4. Ability to get up and down from the floor with minimal assistance;
5. Ability to provide informed consent;
6. No medical contraindication to participation in an exercise program including unstable or active untreated major medical illness (i.e., cardiovascular disease, neurological or neuromuscular diseases, stroke, cancer, etc.);
7. A score of 23 or above on the Montreal Cognitive Assessment;
8. Not currently participating in yoga more than one time per week;
9. Can understand and communicate in English.
10. Willing and bale to provide consent.

Exclusion Criteria:

1. Existing musculoskeletal injury.
2. Severe freezing of gait.
3. Enrolled in another yoga or research program.
4. Unstable or active major medical illness.
5. Answer "Yes" to any questions on the PAR-Q or Elder PAR-Q.
6. Pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Dysfunction | Baseline, Week 19
  The Montreal Cognitive Assessment (MoCA) is a rapid screening instrument for mild cognitive dysfunction. A total possible score is 30 points with a range of 0-30. A score of 26 or above is considered normal.
Change in Executive Function (EF) | Baseline, Week 20.
  The Wisconsin Card Sort task evaluates executive function with correct scores and errors associated with previously used rules known as preservative errors. Scores (t-scores) on the Wisconsin Card Sort task (total error) at study endpoint adjusted for education are min=0 and max=100. Higher scores indicate better outcomes.
Change in Executive Function Measured by Inhibition of Cognitive Inference | Baseline, Week 20
  The Stroop color word test evaluates the participant's ability to inhibit cognitive inference. This is a cognitive domain of executive function and involves the processing of a stimulus where one feature of a previous stimulus may affect the simultaneous processing of a new stimulus. The total score can range from 0 to 100 with higher scores indicating better memory function.
Change in Executive Function as Measured by Changes in Visual Spatial Ability and Task-switching | Baseline, Week 20
  The Trail Making Test Part A & B measures visuospatial abilities, working memory and task switching abilities associated with EF domains. Lower times to completion and fewer errors indicate better performance. Scores for Part A typically can range from 20 to 90 seconds. Scores for Part B can range from 60 seconds to 180 seconds.
Change in Distance Walked in Six Minutes | Baseline, Week 19
  The six-minute walk test measures cardiovascular performance. The test measures how far you can walk in 6 minutes. Scores typically range from 200 to 500 meters in Parkinson's disease (PD) patients.

SECONDARY OUTCOMES:
Changes in body weight | Baseline, Week 19
  Body weight will be measured in kilograms using a Tanita BC-418 bioelectrical impedance scale.
Changes in fat-free mass | Baseline, Week 19
  Fat-free mass will be measured in kilograms using a Tanita BC-418 bioelectrical impedance scale.
Changes in Dynamic Balance | Baseline, Week 19
  The Mini-BESTest measures dynamic balance deficits in persons with mild to moderate PD. The assessment has 14 items. Each item is rated on a 0-2 point scale, where a score of 0 indicates that the participant is unable to complete the task, and a score of 2 indicates normal performance. The score can range from 0 to 28. Higher score indicates better dynamic balance.
Changes in Functional Agility | Baseline, Week 19
  The Timed Up-and-Go measures a participant's ability to rise from a standard chair walk 3 meters, walk around a cone, walk back 3 meters and sit down in the chair. The measure is how long it takes to complete the task. The range of scores is 6.5 seconds to 20.3 seconds. A lower score indicates better agility.
Changes in Reactive Balance Distance | Baseline, Week 19
  Reactive balance testing measures the ability of the participant to maintain balance on a moving platform. The dynamic balance score can range from 1440 centimeters to 0 centimeters, with the lower score indicating better performance.
Changes in Reactive Balance Time | Baseline, Week 19
  Reactive balance testing measures the ability of the participant to maintain balance on a moving platform. The time-on-test score can range from 0-120 seconds with the higher score indicating better performance.
Changes in Perceived Fall Risk | Baseline, Week 19
  The Modified Fall Efficacy Scale measures perceived balance ability and fall risk. The instrument consists of 14 self-report items which are scored on a 10-point Likert based scale. A score of 0 indicates not confident at all and a score of 10 indicates complete confidence. The test can range from 0 to 140.
Changes in Quality of Life | Baseline, Week 19
  The Parkinson's Disease Questionnaire (PDQ-39) measures self-reported quality of life in Parkinson's patients. It has 39 items with an overall score range from 20 to 56 with the lower score indicating better quality of life.
Changes in Motor Function | Baseline, Week 19
  The Unified Parkinson's Disease Rating Scale-III motor scale is an examination of motor dysfunction in Parkinson's disease patients. The score can range from 0 to 108 with the higher score indicating greater dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Max Orovitz Laboratories, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wooten SV, Signorile JF, Desai SS, Paine AK, Mooney K. Yoga meditation (YoMed) and its effect on proprioception and balance function in elders who have fallen: A randomized control study. Complement Ther Med. 2018 Feb;36:129-136. doi: 10.1016/j.ctim.2017.12.010. Epub 2017 Dec 29. PMID 29458919
- [Background] Potiaumpai M, Martins MC, Wong C, Desai T, Rodriguez R, Mooney K, Signorile JF. Difference in muscle activation patterns during high-speed versus standard-speed yoga: A randomized sequence crossover study. Complement Ther Med. 2017 Feb;30:24-29. doi: 10.1016/j.ctim.2016.11.002. Epub 2016 Nov 18. PMID 28137523
- [Background] Potiaumpai M, Martins MC, Rodriguez R, Mooney K, Signorile JF. Differences in energy expenditure during high-speed versus standard-speed yoga: A randomized sequence crossover trial. Complement Ther Med. 2016 Dec;29:169-174. doi: 10.1016/j.ctim.2016.10.002. Epub 2016 Oct 15. PMID 27912943
- [Background] Ni M, Mooney K, Signorile JF. Controlled pilot study of the effects of power yoga in Parkinson's disease. Complement Ther Med. 2016 Apr;25:126-31. doi: 10.1016/j.ctim.2016.01.007. Epub 2016 Feb 10. PMID 27062960
- [Background] Ni M, Signorile JF, Mooney K, Balachandran A, Potiaumpai M, Luca C, Moore JG, Kuenze CM, Eltoukhy M, Perry AC. Comparative Effect of Power Training and High-Speed Yoga on Motor Function in Older Patients With Parkinson Disease. Arch Phys Med Rehabil. 2016 Mar;97(3):345-354.e15. doi: 10.1016/j.apmr.2015.10.095. Epub 2015 Nov 4. PMID 26546987
- [Background] Ni M, Mooney K, Richards L, Balachandran A, Sun M, Harriell K, Potiaumpai M, Signorile JF. Comparative impacts of Tai Chi, balance training, and a specially-designed yoga program on balance in older fallers. Arch Phys Med Rehabil. 2014 Sep;95(9):1620-1628.e30. doi: 10.1016/j.apmr.2014.04.022. Epub 2014 May 14. PMID 24835753
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886